CLINICAL TRIAL: NCT05525507
Title: A Single-armed, Unblinded, Non-randomized Feasibility Study of Hematopoietic Stem Cell Infusion Following a Conditioning Regimen of Total Lymphoid Irradiation (TLI) and Anti-thymocyte Globulin (ATG) in Patients With a Pre-existing, Well-functioning HLA-matched Kidney Transplant
Brief Title: Delayed Immunological Tolerance in Patients With Well-functioning Pre-existing HLA-matched Kidney Transplants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey Veale, MD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Delayed Tolerance
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: End Stage Kidney Disease; Immunological Tolerance; Kidney Transplant Failure and Rejection; Chronic Kidney Diseases
Keywords: immunological tolerance; kidney transplant; tolerance; end stage kidney disease; end stage renal disease; chronic kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Rejection, Psychology; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immune tolerance in HLA-identical kidney transplant recipient (Experimental): We seek to establish immunological tolerance in patients with a pre-existing, well- functioning kidney transplant from an HLA-identical donor. Patients will undergo conditioning with TLI and ATG, followed by infusion of hematopoietic stem cells from the same donor . We will evaluate whether recipients can be withdrawn from immunosuppressive drugs without compromising allograft function. At serial time points, graft function will be monitored, and chimerism will be measured. Weaning of tacrolimus will begin at 6 months, with a goal of drug discontinuation within 12 months if the following conditions are met: (1) chimerism (defined as ≥1% donor type cells among the T cells, B cells, NK cells, and granulocytes) is detectable for at least 180 days, (2) stable graft function (defined as eGFR >30 mL/min and no greater than sustained 30% change over 3 months from baseline) without clinical rejection episodes is maintained, and (3) no evidence of graft vs. host disease (GVHD).
  Interventions: Combination Product: Conditioning and Stem cell infusion

INTERVENTIONS:
Combination Product: Conditioning and Stem cell infusion — Patients will undergo a conditioning with TLI and ATG, followed by infusion of hematopoietic stem cells from the same HLA-identical donor that provided the original kidney

SUMMARY:
The study seeks to determine if patients with a pre-existing, well-functioning kidney transplant from a HLA-identical living donor can be withdrawn from immunosuppressive medications without compromising allograft function through hematopoietic stem cell (HPSC) infusion from the same donor. HPSC infusion will be preceded by a conditioning regimen of total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (rATG).

DETAILED DESCRIPTION:
Immunological tolerance through combined kidney and HPSC transplant has been demonstrated at few centers of excellence within the United States. The ultimate aim of these protocols is to liberate patients from lifelong immunosuppression. Thus far, protocols have been limited to HLA-identical donor recipient pairs, undergoing simultaneous kidney transplant and HPSC infusion. In all protocols, the recipient undergoes a conditioning regimen to optimize engraftment. Our protocol employs a conditioning regimen of TLI and ATG.

There are many more patients with pre-existing well-functioning HLA-identical kidney transplants than those who present de novo for participation in tolerance trials. Despite this, post hoc tolerance induction through HPSC infusion in patients with a pre-existing kidney transplant has not yet been performed. Given the demonstrated success of tolerance protocols in simultaneous haploidentical kidney and HPSC transplant, the next logical step is to demonstrate that tolerance can be induced in the much greater subset of patients with pre-existing kidney transplants.

This study employs an established protocol for immunological tolerance induction in patients with a pre-existing, well- functioning kidney transplant from their haploidentical donor. These patients will undergo a conditioning with TLI and ATG, followed by infusion of HPSC from the same HLA-identical donor that provided the original kidney. The Investigators call this process "retroactive tolerance induction."

The investigators will evaluate whether recipients can be withdrawn from immunosuppressive drugs without compromising allograft function. At serial time points, (1) graft function will be monitored, and (2) chimerism will be measured in recipient whole blood and white blood cell subsets. Weaning of tacrolimus will begin at 6 months, with a goal of drug discontinuation within 12 months if the following conditions are met: (1) chimerism (defined as ≥1% donor type cells among the T cells, B cells, NK cells, and granulocytes) is detectable for at least 180 days after CD34+ and CD3+ cell infusion, (2) stable graft function (defined as eGFR >30 mL/min and no greater than sustained 30% change over 3 months from baseline) without clinical rejection episodes is maintained, and (3) there is no evidence of graft vs. host disease (GVHD).

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Males and females ages 18 years and older with a pre- existing kidney transplant from an HLA-matched living donor.
2. Pre-existing living kidney transplant must be within 3 months to 5 years from date of scheduled HPSC infusion.
3. No history of rejection with current HLA matched kidney transplant.
4. Recipient is without post-transplant major complications, including de novo malignancy, active infection or rejection.
5. Stable renal function determined per investigator discretion.
6. Agreement to participate in the study and ability to give informed consent.
7. Meets institutional criteria for HSPC infusion.
8. Resides or is willing to stay within 3 hours distance from UCLA Medical Center by ground transportation for the first three to six months of the trial at the physician's discretion.
9. No known contraindication to administration of rATG or radiation.
10. If participant is a female of reproductive potential (i.e., no documented absence of ovaries or uterus, history of tubal ligation, or post-menopausal status) participant must be confirmed not pregnant by a serum or urine pregnancy test) and must agree to practice a reliable form of contraception including hormonal treatments, barrier methods or intrauterine device for at least 12 months post-transplant.
11. Karnofsky Performance Score (KPS) ≥ 70.
12. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 40% by MUGA (Multi Gated Acquisition) scan or echocardiogram.
13. Adequate liver function defined as total bilirubin ≤ 1.5 times the upper limit of normal and AST/ALT ≤ 2.0 times the upper limit of normal.
14. Adequate social support based on evaluation by the UCLA bone marrow and/or renal transplant team.

Recipient Exclusion Criteria:

1. Donor is identical twin.
2. Major ABO incompatibility with donor
3. Positive HLA Donor-Specific Antibody (DSA)
4. History of multi-organ transplantation
5. History of rejection with current HLA-matched kidney transplant
6. Known allergy to rabbit proteins
7. History of post-transplant major complications, including de novo malignancy, active/chronic infection or rejection, with the exception of low risk, early-stage malignancy with

   ≥90% 5-year survival not receiving chemotherapy or immunotherapy and non-melanomatous skin cancer.
8. History of active malignancy within the past 5 years with the exception:

   1. Low risk cancer on active surveillance
   2. Malignancy treated with curative intent with no known active disease >2 years before the first dose of study treatment and of low potential risk for recurrence
   3. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   4. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ, and DCIS)
9. Worsening renal functioning over preceding 3-month interval determined per investigator discretion.
10. Pregnant (confirmed by urine or serum pregnancy test) or lactating.
11. Leukopenia (with a white blood cell count < 3,000/µL) or thrombocytopenia (with a platelet count < 70,000/µL).
12. EBV, CMV and BK PCR negative at time of HPSC infusion is preferred, but if they have had a history of + CMV/BK PCR, it should be resolved by 3 months.
13. Active bacterial, fungal, mycobacterial, or viral infection (including active hepatitis B and/or C).
14. Seropositivity for HIV 1 or 2 by 4th generation serum antibody/antigen testing, or HTLV I or II by serum antibody testing.
15. Renal disease with high risk of recurrence (i.e., focal segmental glomerulosclerosis).
16. Advanced hepatic fibrosis or cirrhosis secondary to hepatitis B and/or C diagnosis.
17. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia; active extra-renal autoimmune disease requiring immunosuppression.
18. Active extra-renal autoimmune disease requiring immunosuppression.
19. Neuropsychiatric illness that precludes the ability to give informed consent and/or places the participant as high risk for non-compliance with the safety monitoring requirements of the study.
20. May not have received other immunomodulatory agents, including but not limited to tumor necrosis factor inhibitors within six months of the study treatment. Use of corticosteroids prescribed for a time-limited indication (</= 4 weeks) and stopped at least 4 weeks before the kidney transplant is acceptable.
21. May not have received immunotherapy drugs such as immune checkpoint inhibitors (e.g. pembrolizumab, nivolumab, and ipilimumab), tumor necrosis factor inhibitors, rituximab, and interleukin-2 within six months of the study treatment.
22. Current or active abuse of alcohol and/or drugs within last 6 months.
23. Body Mass Index (BMI) ≥ 40.

Donor Inclusion Criteria:

1. HLA-matched sibling on high-resolution HLA typing who

   a. is ≥18 years of age.
2. Must meet institutional criteria for HSPC transplant donation.
3. Medically fit to tolerate peripheral blood apheresis, including weighing ≥110 pounds, hemoglobin ≥11, white blood cell count ≥ 3,000/µL, and platelets ≥ 100,000/µL.
4. Serum creatinine as expected post-kidney donation and coagulation parameter studies; or, if abnormal, the changes are not considered clinically significant.

Donor exclusion criteria:

1. Recipient is identical twin.
2. Major ABO incompatibility with recipient.
3. Medically unfit to tolerate peripheral blood apheresis (e.g. small body size, poor vascular access, not a suitable candidate for placement of a central catheter).
4. Pregnant (confirmed by urine or serum pregnancy test) or lactating.
5. Seropositivity for HIV 1 or 2 by 4th generation serum antibody/antigen testing, HTLV I or II by serum antibody testing
6. Active West Nile Virus infection.
7. Active bacterial, fungal, mycobacterial or viral infection (including active hepatitis B and/or C).
8. Psychiatric, addictive, neurological, or other disorder that compromises ability to give true informed consent for participation in this study.
9. History of active malignancy within the past 5 years with the exception:

   1. Low risk cancer on active surveillance
   2. Malignancy treated with curative intent with no known active disease >2 years before the first dose of study treatment and of low potential risk for recurrence
   3. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   4. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ, and DCIS)
10. No use of oral anticoagulants 2 days prior to apheresis. Note: Use of aspirin and non-steroidal anti-inflammatory drugs, for pain and inflammation management purposes, are permitted to enroll in the study, but these drugs must be stopped 7 days prior to apheresis, however subjects who are taking aspirin for its anti- platelet/anti-thrombotic effect, are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of successful discontinuation of immunosuppression | 12 months
  To determine whether patients with pre-existing kidney transplants from a haploidentical living donor can be withdrawn from immunosuppressive drugs while maintaining stable graft function within 12 months of hematopoietic stem cell infusion from the same HLA-identical living donor, preceded by conditioning with TLI and ATG.

SECONDARY OUTCOMES:
Incidence of allograft rejection | 48 months
  To determine the percentage of subjects with graft rejection within 48 months post-HPSC infusion defined as (1) meets Banff criteria for rejection on biopsy performed to confirm clinical suspicion of rejection or (2) clinical suspicion of rejection demonstrating response to corticosteroids in absence of biopsy when confirmatory biopsy contraindicated or declined.
Graft survival | 24 months
  To determine graft survival within the first 24 months post-HPSC infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Veale, MD, Principal Investigator — Professor of Urology
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No